CLINICAL TRIAL: NCT07237555
Title: Comparison of the Likelihood of Side Effects Between Surgical Methods in Patients With Severe Stage Glaucoma
Brief Title: CVL Risk After Severe Glaucoma Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Wungrak choi, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2024-0364
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Severe-stage Glaucoma (Mean Deviation ≤ -20 dB)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 231 eyes that underwent trabeculectomy for severe-stage glaucoma
- Group 2: 292 eyes that underwent Ahmed glaucoma valve implantation for severe-stage glaucoma

SUMMARY:
This retrospective cohort study analyzes risk factors for central visual loss (CVL) after severe-stage glaucoma surgery. The primary hypothesis is that 1) visual prognosis is determined primarily by early postoperative intraocular pressure (IOP) stability rather than surgical choice, and 2) the nature of risk (hypotony vs hypertension) is modified by baseline visual reserve. We analyzed outcomes in 523 patients with severe-stage glaucoma who underwent trabeculectomy or Ahmed glaucoma valve (AGV) implantation, focusing on the dichotomous risk profile stratified by baseline visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who underwent trabeculectomy or Ahmed glaucoma valve implantation at Yonsei Medical Center between January 2005 and October 2024.

  2. Glaucoma patients who underwent static quantitative perimetry (visual field test) before and after surgery.

  3. Patients with a preoperative Mean Deviation (MD) of ≤ -20 dB.

Exclusion Criteria:

* 1. Patients who were unable to undergo visual field testing due to poor preoperative visual acuity.

  2. Patients with central visual field defects caused by retinal or neurological diseases other than glaucoma.

  3. Patients with false-positive or false-negative responses ≥33% on visual field testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe-stage glaucoma who underwent trabeculectomy or Ahmed glaucoma valve implantation at Gangnam Severance Hospital, Yonsei University College of Medicine, between January 2005 and October 2023, with at least 1-year follow-up data available.
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Central Visual Loss (CVL) at 3 months postoperatively | At 3 months postoperatively
  Central visual loss defined as any of the following at 3 months postoperatively: (i) best-corrected visual acuity (BCVA) ≤ 20/200; (ii) decrease of ≥ 4 Snellen lines from baseline; or (iii) further deterioration of BCVA in eyes with preoperative BCVA ≤ 20/200.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severacne Hospital, Seoul, South Korea

REFERENCES:
- [Background] Mills RP, Budenz DL, Lee PP, Noecker RJ, Walt JG, Siegartel LR, Evans SJ, Doyle JJ. Categorizing the stage of glaucoma from pre-diagnosis to end-stage disease. Am J Ophthalmol. 2006 Jan;141(1):24-30. doi: 10.1016/j.ajo.2005.07.044. PMID 16386972
- [Background] Bai J, Smock SL, Jackson GR Jr, MacIsaac KD, Huang Y, Mankus C, Oldach J, Roberts B, Ma YL, Klappenbach JA, Crackower MA, Alves SE, Hayden PJ. Phenotypic responses of differentiated asthmatic human airway epithelial cultures to rhinovirus. PLoS One. 2015 Feb 23;10(2):e0118286. doi: 10.1371/journal.pone.0118286. eCollection 2015. PMID 25706956
- [Background] Zhu S, Li ZW, Zhao H. Patchy micelles based on coassembly of block copolymer chains and block copolymer brushes on silica particles. Langmuir. 2015 Apr 14;31(14):4129-36. doi: 10.1021/acs.langmuir.5b00526. Epub 2015 Apr 1. PMID 25811763
- [Background] Pernas M, Garcia-Casado G, Rojo E, Solano R, Sanchez-Serrano JJ. A protein phosphatase 2A catalytic subunit is a negative regulator of abscisic acid signalling. Plant J. 2007 Sep;51(5):763-78. doi: 10.1111/j.1365-313X.2007.03179.x. Epub 2007 Jul 7. PMID 17617176
- [Background] Lambiase A, Micera A, Sacchetti M, Cortes M, Mantelli F, Bonini S. Alterations of tear neuromediators in dry eye disease. Arch Ophthalmol. 2011 Aug;129(8):981-6. doi: 10.1001/archophthalmol.2011.200. PMID 21825181